CLINICAL TRIAL: NCT03243500
Title: Efficacy and Safety of Low Dose Atracurium Added to Lidocaine, Bupivacaine and Hyaluronidase Mixture in Percaruncular Peribulbar Anesthesia for High Myopes Undergoing Phacoemulsification: A Randomized Controlled Trial.
Brief Title: Efficacy and Safety of Adding Atracurium to Percaruncular Block for High Myopes Undergoing Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Assistant Lecturer - Anesthesia, pain management and surgical ICU department, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 14/9/2014
Record Dates: First submitted 2017-08-02; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Quality of Ocular Akinesia (Onset and Duration)
Keywords: atracurium; high myopes; percaruncular; phacoemulsification; medial canthal; ophthalmic regional anesthesia
MeSH Terms: interventions — Atracurium; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Sham Comparator): 2.5 ml of lidocaine 2% 2.5 ml of bupivacaine 0.5% hyaluronidase powder 15 IU/ml
  1 ml normal saline to make a total volume of 6 ml from which the patient received 5-6 ml through percaruncular peribulbar injection.
  Interventions: Drug: Lidocaine 2%; Drug: Bupivacaine 0.5%; Drug: hyaluronidase powder; Procedure: per-caruncular peribulbar injection
- Group A (Active Comparator): 5 mg atracurium 2.5 ml of lidocaine 2% 2.5 ml of bupivacaine 0.5% hyaluronidase 15 IU/ml
  1 ml normal saline to make a total volume of 6 ml from which the patient received 5-6 ml through percaruncular peribulbar injection.
  Interventions: Drug: Atracurium; Drug: Lidocaine 2%; Drug: Bupivacaine 0.5%; Drug: hyaluronidase powder; Procedure: per-caruncular peribulbar injection

INTERVENTIONS:
Drug: Atracurium — 5mg in 1 ml normal saline
  Other Names: atracurium besylate
  Arms: Group A
Drug: Lidocaine 2%
  Other Names: lidocaine hydrochloride 2%
Drug: Bupivacaine 0.5%
  Other Names: Sunnypivacaine 0.5%
Drug: hyaluronidase powder — 1500 iu powder diluted in 2 vial lidocaine 20 ml resulting 37.5 IU/ml lidocaine and 93.7 / 2.5 ml lidocaine or 15.6 IU/ml of the 6 ml solution
  Other Names: Omnidase 1500iu Injection
Procedure: per-caruncular peribulbar injection — The patient will lie in a supine position and the eyes are in the neutral position. The needle (25 Gauge (G), 25 mm) insertion point will be just medial to the caruncle, directly perpendicular to the face and parallel to the medial orbital wall to 15-20 mm depth. After negative aspiration the already chosen local anesthetic mixture will be injected slowly. During injection, the globe will be palpated with one finger and tension in the lids will be tested frequently, if the lids become tense or if the tension is felt to rise in the globe, the injection will be stopped. After injection, external compression with Honan balloon inflated to 20-30 mm Hg will be applied for 10 minutes and will be removed every 2 minutes to test akinesia and anesthesia
  Other Names: medial canthal block

SUMMARY:
There are several local anesthetic techniques available for cataract surgery and the choice depends on patient, surgical and operator factors. The eyes of patients with axial myopia (the eye globe is abnormally elongated) have thin wall (sclera), limited space for needle insertion for local anesthetic injection between the globe and the orbit and out-pouching of the back of the eye (staphyloma). These factors increased the risk of perforation following conventional needle techniques of eye block The current study technique is per-caruncular injection (the needle insertion site is between the nasal side of the globe and bony orbit) which may provide a safer alternative to the conventional needle techniques for myopic patients. The space of injection is devoid of blood vessels moreover, myopic staphylomata are infrequently located on the nasal side of the globe.

Local injection of muscle relaxant added to local anesthetic solution may provide earlier onset of eye muscle paralysis thus earlier onset of favorable surgical condition than local anesthetic solution alone.

The current study will demonstrate the effect of adding low dose atracurium (a muscle relaxant) to local anesthetic mixture in providing early onset of eye muscle paralysis and favorable surgical condition in per-caruncular technique of eye block in high myopes undergoing cataract surgery.

DETAILED DESCRIPTION:
In the current study, it is hypothesized that adding low dose atracurium to lidocaine, bupivacaine and hyaluronidase mixture would provide an early onset of akinesia and favorable surgical condition in per-caruncular peribulbar anesthesia for high myopes undergoing phacoemulsification Initially, informed consents from the eligible patients will be obtained. Preoperatively, the axial length of the enrolled patients will be measured by ultrasound biometry and the presence of staphyloma was identified by B-scan.

In the preparation room, the intravenous (IV) cannula will be placed. Anxious patients will be given midazolam intravenously (titrated to response according to patient's age and associated medical condition).

In the operating room, standard monitoring of pulse oximetry, electrocardiography (ECG) and noninvasive arterial blood pressure will be commenced. The O2 will be administered at 2 ml/minutes by the nasal O2 cannula. Drugs and equipment for resuscitation will be checked before initiation of the procedure.

Local anesthetic eye drops (benoxinate 0.4%) will be instilled in the eye to be operated upon three times separated by one minute interval.

The patient will lie in a supine position and will be asked to look directly ahead focusing on a fixed point on the ceiling, so that the eyes are in the neutral position. A per-caruncular will be given using a 25 Gauge (G), 25 mm needle. The needle insertion point will be just medial to the caruncle with the needle passing directly perpendicular to the face and parallel to the medial orbital wall to 15-20 mm depth. , After negative aspiration the already chosen local anesthetic mixture will be injected slowly. During injection, the globe will be palpated with one finger and tension in the lids will be tested frequently, if the lids become tense or if the tension is felt to rise in the globe, the injection will be stopped. After injection, external compression with Honan balloon inflated to 20-30 mm Hg will be applied for 10 minutes and will be removed every 2 minutes to test akinesia and anesthesia.

The following will be recorded:

* Age.
* Sex.
* ASA physical status.
* Axial length.
* Blood pressure, heart rate (baseline, 5 minutes after local anesthetic injection, 5 minutes after the beginning of the operation)
* peripheral O2 saturation (SpO2) (baseline and 5 minutes after local anesthetic injection) were recorded.
* The beginning of motor blockade (ocular movement score [OMS]≤6) and onset time of globe akinesia (OMS≤2)will be recorded. Moreover, the OMS will be assessed at the end of the surgery and then every 30 minutes post-operative till regaining full ocular movement to determine the duration akinesia.
* The time to eyelid movement score of ≤1 will be recorded. If, after 10 minutes the block is inadequate a 3-4 ml supplementation of lidocaine 2% by the same technique will be given. If the block is still inadequate, it will be considered a failure and excluded from the study. When the block is considered a failure the patient will receive either supplemental inferotemporal injection (if ultrasound excluded presence of posterior staphyloma), topical anesthesia, intravascular fentanyl 50 mcg or general anesthesia according to the patient condition.

After adequate analgesia (loss of sensation to touch by a small cotton wool) and akinesia (OMS≤2), the surgeon was allowed to start the surgery.

* The need for supplementation and total volume of local anesthetic mixture will be recorded.
* Time to adequate surgical anesthesia will be noted defined as the presence of corneal anesthesia together with ocular movement score ≤2.
* Pain will be assessed by direct questioning using a 3 point scoring system:

(No pain = 0, discomfort = 1, pain = 2) throughout the operation. If the patient score is 1 or more, reassurance and or 50 mcg fentanyl IV will be given.

* The occurrence of complication (Retrobulbar hemorrhage, Globe penetration, Optic nerve damage, Local anesthetic toxicity, Muscle palsies, Chemosis, or side effect of the muscle relaxant e.g. local hyperemia) will be recorded.
* The duration of the procedure will be recorded.
* Surgeon satisfaction will be assessed at the end of surgical procedure by using a three-point scale: 0 = not satisfied, 1 =moderately satisfied, 2 = satisfied.

The data collector (also the administrator of the block) will record the data in a pre-printed data sheet with abbreviations and each variable is explained. Also in the data sheet, principle investigator number and e-mail for communication will be present. The collected data will be then revised and registered to an electronic form for later statistical analysis.

Sample size Based on a two-sided alpha of 0.05, 95% power, and a clinically relevant difference in time of onset of akinesia at least 3 minutes, a minimum of 74 patients will be required for the conduct of the study (MedCalc®version12.7.1.0- 64-bit). Eight patients will be added to compensate for dropouts.

82 patients will be randomly allocated into 2 groups: Statistical analysis Statistical analysis will be performed using S-Plus Statistical Software (SPSS) for Windows (version 20.0, SPSS Inc. Chicago, Illinois). All variables will be tested for normality using Kolmogorov-Smirnov test; if the test is significant, non-normality will be accepted. Otherwise double-checking using graphs, skewness and kurtosis will be required to confirm normality.

Continuous variables will be presented as mean ± standard deviation when normality of distribution assumptions are satisfied. If not, it will be presented as median and range. categorical variables will be presented as numbers and percentages. Quantitative variables will be compared using two-tailed unpaired student t- test, and qualitative variables will be compared using Fisher's exact test. P value of < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* high myopia (axial length 26mm or more)

Exclusion Criteria:

* Pregnant patients.
* ASA physical status >III.
* Axial length less than 26 mm.
* Contraindication of regional anesthesia:

Absolute contraindications: Patient refusal to participate in the study, Local anesthetic allergy and Infection/marked orbital inflammation or, Relative contraindications: unable to lie flat for a sufficient length of time, Confusion or psychiatric illness, communication difficulties, bleeding diathesis or taking anticoagulants, Previous scleral buckling or space-occupying lesions within the orbit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
assessing the quality of akinesia (onset and duration) of low dose atracurium added to lidocaine, bupivacaine and hyaluronidase mixture in Percaruncular peribulbar block | from onset of ocular akinesia up to 24 hours postoperatively
  This will be achieve by assessing ocular movement score (OMS) every 2 minutes by asking the patient to move his/her eye in four directions; up, down, medially and laterally and the movement in each direction is given a score from 0 to 2 as follows: movement more than 2 mm will be given a score of 2, 1-2 mm movement will be given a score of 1 and no movement will be given a score of 0. A total Score of 2 or less will be considered adequate akinesia for surgery.
  Also, eyelid movement score will be assessed by asking the patient to open his/her eye widely followed by squeezing them maximally. A full movement will be given a score of 2, the flickering will be given a score of 1 and no movement will be given a score of 0.

CONTACTS AND LOCATIONS:
Overall Officials: nazmy e seif, md, Study Director — lecturer at Anesthesia, Pain Management and Surgical ICU Department, Cairo University, Egypt; ashraf m Amin, md, Study Chair — professor at Anesthesia, Pain Management and Surgical ICU Department, Cairo University, Egypt; Mahmoud m Soliman, md, Study Director — MD and professor at Ophthalmology Department, Cairo University, Egypt.; maha m Ismail, md, Study Director — MD and assistant professor at Anesthesia, Pain Management and Surgical ICU Department, Cairo University, Egypt; Maha M Ahmad, md, Principal Investigator — assistant lecturer at Anesthesia, Pain Management and Surgical ICU Department, Cairo University, Egypt.
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided